CLINICAL TRIAL: NCT05650528
Title: Single-center, Randomised, Double-blind, Placebo-controlled Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile of Single- and Multiple-dose Ascending Oral QG101-23-0 Capsules in Healthy Subjects
Brief Title: QG101-23-0 Capsules SAD and MAD Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amckaus PTY LTD. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Aom0315-ACT-01
Record Dates: First submitted 2022-11-29; First posted 2022-12-14 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part A (Experimental): Six single-ascending dose levels (Cohort A1\Cohort A2\Cohort A3\Cohort A4\Cohort A5\Cohort A6) of SAD QG101-23-0 capsules (n=6) or placebo (n=2)
  Interventions: Drug: QG101-23-0 capsules; Drug: Placebo
- Part B (Experimental): Three multiple-ascending dose levels (Cohort B1\Cohort B2\Cohort B3) of MAD QG101-23-0 capsules (n=6) or placebo (n=2)
  Interventions: Drug: QG101-23-0 capsules; Drug: Placebo
- Part C (Experimental): Cohort A3 Group 1 (n=8) and Group 2 (n=6, additional recruitment) participated in the food effect study. The subjects took QG101-23-0 capsules while under fasting or fed condition.
  Interventions: Drug: QG101-23-0 capsules; Drug: Placebo

INTERVENTIONS:
Drug: QG101-23-0 capsules — Single and Multiple Dose for oral
Drug: Placebo — Single and Multiple Dose for oral

SUMMARY:
The study will consist of three parts: a single-dose ascending (SAD) phase (Part A) enrolling a total of five ~ six cohorts of healthy participants, a multiple-dose ascending (MAD) phase (Part B) enrolling 3 cohorts of healthy participants, and a food effect study (Part C).

DETAILED DESCRIPTION:
This study is a single-center, randomized, double-blind and placebo-controlled trial. Healthy subjects will receive single- and multiple-dose administration through oral of different doses of QG101-23-0 capsules to evaluate its safety, tolerability and pharmacokinetics profile.

ELIGIBILITY:
Inclusion Criteria：

Subjects must satisfy all the following criteria at the Screening visit and Check-in unless otherwise stated:

1. Males or females, between 18 and 55 years of age, inclusive.
2. Body weight is ≥ 50.0 kg for male subjects and ≥ 45.0 kg for female subjects, with a body mass index (BMI) of 18-32 kg / m2 (inclusive).
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs measurements, and clinical laboratory evaluations at Screening and Check-in as assessed by the Investigator (or designee), as applicable. Resting heart rate ≥ 45 bpm and ≤ 100 bpm at Screening.
4. Male subjects must agree to refrain from sperm donation from the time of signing the informed consent form until 90 days after the last dosing and females should refrain from ova donation from the time of signing the informed consent form until 30 days after the last dosing. As detailed in Appendix 2.
5. Females will not be pregnant or lactating, female subjects with a negative blood pregnancy test during the Screening period and a negative urine pregnancy test at Check-in, and male and female of childbearing potential having taken effective contraceptive measures at least from the date of signing the informed consent form and should agree to continue to use effective contraceptive measures from the date of signing the informed consent form until 90 days after the last dosing for males and 30 days after the last dosing for females. Males with vasectomy at least 90 days prior to the Screening visit must have documentation confirming Azoospermia or use other contraceptives. As detailed in Appendix 2.
6. Females of nonchildbearing potential defined as permanently sterile (i.e., due to hysterectomy, bilateral salpingectomy, and/or bilateral oophorectomy; at least 3 months between sterlization date and screening date) or postmenopausal (defined as at least 12 months post cessation of menses without an alternative medical cause and follicle-stimulating hormone [FSH] level ≥ 30 IU/L). As detailed in Appendix 2.
7. Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions.

Exclusion Criteria：

Subjects will be excluded from the study if they satisfy any of the following criteria at the Screening visit and Check-in unless otherwise stated:

1. Significant history or clinical manifestation of any metabolic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, acute or chronic infectious diseases and malignancies, as determined by the Investigator (or designee).
2. History of hereditary bleeding disorders, coagulation disorders, non-traumatic bleeding requiring treatment, or thromboembolism; or currently have any disease that can cause bleeding (including coagulation disorder, thrombocytopenia [platelet count < 150×109/L] and prothrombin time-international normalised ratio > 1.5);
3. Acute and chronic liver disease or serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 1.5 × the upper limit of normal at Screening or Check-in;
4. History of acute and chronic kidney disease including acute and chronic renal insufficiency. Or impaired renal function defined by creatinine clearance (calculated using the Cockcroft-Gault equation) < 90 mL/min at Screening or Check-in; See Appendix 3 Formulas Used in the Study.
5. Abnormal blood pressure (defined as systolic blood pressure > 145 mmHg or < 90 mmHg, diastolic blood pressure > 90 mmHg or < 50 mmHg) at Screening or Check-in;
6. History of clinically significant hypersensitivity, any intolerance, or any anaphylaxis to any drug compound including any components of the study drug capsules, such as lactose, hydroxypropyl methylcellulose, magnesium stearate, food, or other substance, unless approved by the Investigator (or designee).
7. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), and/or positive human immunodeficiency virus (HIV) test at Screening. Participants with previously treated HCV and hence HCV Ab positive may be included if a subsequent HCV RNA test is negative.
8. Any of the following on the ECG at Screening and Check-in (Day -1).

   1. ECG is abnormal and clinically significant, or the corrected QTc interval (QTc is calculated by Fridericia correction formula: QTc = QT/ [RR ^ 0.33]) > 450 msec (male) or > 470 msec (female) is confirmed by repeat measurement at least two times. See Appendix 3 Formulas Used in the Study.
   2. QRS duration > 120 msec, confirmed by repeat measurement at least two times.
   3. PR interval > 220 msec, confirmed by repeat measurement at least two times.
   4. Findings which would make QTc measurements difficult or QTc data uninterpretable.
   5. History of additional risk factors for torsades de pointes (e.g., heart failure, hypokalaemia, family history of long QT syndrome).
   6. Abnormal QRS or ST segment indicates a clinically significant abnormality of myocardia, e.g., cardiomyopathy, cardiac ischaemia or myocardial infarction, etc.
9. History of stomach or intestinal surgery or resection, vagotomy, or any surgery (uncomplicated appendectomy and hernia repair will be allowed, but not cholecystectomy) or adverse syndromes (such as Crohn's disease, Irritable Bowel Syndrome , chronic pancreatitis or congenital nonhaemolytic hyperbilirubinemia [e.g., suspicion of Gilbert's syndrome based on total and direct bilirubin, the subjects with total or direct or indirect bilirubin > 35%× the upper limit of normal at Screening or Check-in]) that would potentially alter gastrointestinal peristalsis, pH, absorption and/or excretion of orally administered drugs.
10. Pregnant or lactating females or females of childbearing potential and males are unwilling to take effective contraceptive measures.
11. Having foods and beverages containing poppy seeds, grapefruit and orange including Seville oranges or wine containing extracts from the above fruits within 3 days prior to Check-in until the follow-up visit.
12. Use or intend to use any medications / products including any prescription or over-the-counter drugs known to alter drug absorption, metabolism, or elimination processes, including vitamin therapy, minerals, and phytotherapeutic / traditional Chinese medicine such as St. John's wort /plant-derived preparations, within 30 days prior to the first dose of study medication until completion of the follow-up visit, unless deemed acceptable by the Investigator (or designee).
13. Having lost blood or donated blood 500 mL or more, within 56 days prior to Screening. Receipt of blood products within 60 days prior to Check-in. The Participants who plan to donate blood from the Screening to 56 days after the follow-up visit.
14. Participation in a clinical study involving administration of an investigational drug or having received any vaccines (including any new investigational vaccines and any approved vaccines such as influenza or COVID-19 vaccines) or a biological product within 30 days (or within five half-lives of the test drug) prior to dosing.
15. History of drug/chemical abuse or substance abuse; Regular consumption of the amount of alcohol (in an Australian standard drink) of more than two standard drinks per day or 14 standard drinks per week within 6 months prior to your admission to the clinical unit (One standard drink is equivalent to 10 grams of alcohol: approximately 285 mL full-strength beer or cider [4.9%], 375 mL mid-strength beer [3.5%], 425 mL light- strength beer [2.7%], 100 mL wine or 30 mL shot of 40% spirit). A positive alcohol breath test at Screening or Day -1, or inability to abstain from alcohol during the study (Within 3 days prior to Check-in until the follow-up visit); Urine drugs of abuse testing as detailed in Appendix 4.
16. Positive alcohol breath test result or positive urine drug screen at Screening or Check-in. Urine drugs of abuse testing as detailed in Appendix 4.
17. History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection at Check-in.
18. Smoke more than five cigarettes per day within 30 days prior to dosing (Day 1) or inability to abstain from tobacco- or nicotine-containing products during the study (Within 3 days prior to Check-in until the check-out) or positive at Screening or Check-in for any other reason.
19. Poor peripheral venous access.
20. History of constipation or the inability to maintain regular bowel movements for the subjects of Cohort A3 within 3 months before administration.
21. In addition to the above, subject who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of single-dose ascending of oral QG101-23-0 capsules in healthy subjects | Day1-8 (SAD)
  Safety will be assessed by the number, severity and type of adverse events, including changes in clinical laboratory evaluations (e.g., Hematology, urinalysis, blood biochemistry, coagulation), vital signs (blood pressure, pulse rate, tympanic thermometers temperature and respiratory rate), ECGs (e.g., QTc interval, QRS duration, PR interval) and physical examinations
The safety and tolerability of multiple-dose ascending oral QG101-23-0 capsules in healthy subjects | Day1-15 (MAD)
  Safety will be assessed by the number, severity and type of adverse events, including changes in clinical laboratory evaluations (e.g., Hematology, urinalysis, blood biochemistry, coagulation), vital signs (blood pressure, pulse rate, tympanic thermometers temperature and respiratory rate), ECGs (e.g., QTc interval, QRS duration, PR interval) and physical examinations

SECONDARY OUTCOMES:
Maximum observed concentration（Cmax） | Day1-8 (SAD)
  Pharmacokinetics
Time of Cmax（Tmax） | Day1-8 (SAD)
  Pharmacokinetics
Area under the concentration-time curve (AUC) from time 0 to the time of the last quantifiable concentration（AUC0-t） | Day1-8 (SAD)
  Pharmacokinetics
AUC from time 0 to 12 hours（AUC0-12） | Day1-8 (SAD)
  Pharmacokinetics
AUC from time 0 to 24 hours（AUC0-24） | Day1-8 (SAD)
  Pharmacokinetics
AUC extrapolated from time 0 to infinity（AUC0-∞） | Day1-8 (SAD)
  Pharmacokinetics
Apparent terminal elimination half-life （t1/2） | Day1-8 (SAD)
  Pharmacokinetics
Apparent distribution volume corrected for bioavailability（Vd/F） | Day1-8 (SAD)
  Pharmacokinetics
Apparent volume of distribution at steady-state (Vss) | Day1-8 (SAD)
  Pharmacokinetics
Apparent terminal elimination rate constant (λz) | Day1-8 (SAD)
  Pharmacokinetics
Mean residence time (MRT) | Day1-8 (SAD)
  Pharmacokinetics
Apparent total clearance (CL) | Day1-8 (SAD)
  Pharmacokinetics
Observed maximum concentration at steady state (Cmax,ss) | Day1-15 (MAD)
  Pharmacokinetics
Observed minimum concentration at steady state (Cmin,ss) | Day1-15 (MAD)
  Pharmacokinetics
Time of Cmax at steady state (Tmax,ss) | Day1-15 (MAD)
  Pharmacokinetics
Average Concentration at steady state (Cav,ss) | Day1-15 (MAD)
  Pharmacokinetics
Time of observed minimum concentration at steady state (Tmin,ss) | Day1-15 (MAD)
  Pharmacokinetics
After steady state, the interval from 0 point of one administration to administration τ Area under the plasma concentration - time curve (AUC0-τ，ss) | Day1-15 (MAD)
  Pharmacokinetics
After steady state, the area under the blood concentration - time curve from 0 point of one administration to infinity （AUC0-∞，ss） | Day1-15 (MAD)
  Pharmacokinetics
Area under the concentration-time curve from time 0 to the end of the dosing interval (AUC0-tau) | Day1-15 (MAD)
  Pharmacokinetics
Area under the concentration-time curve from time 0 extrapolated to infinity (AUC0-inf) | Day1-15 (MAD)
  Pharmacokinetics
Apparent terminal elimination half-life (t1/2) | Day1-15 (MAD)
  Pharmacokinetics
CL for bioavailability at steady state (CL/F, ss) | Day1-15 (MAD)
  Pharmacokinetics
Vd/F at steady state (Vd/F, ss) | Day1-15 (MAD)
  Pharmacokinetics
Mean residence time (MRT) | Day1-15 (MAD)
  Pharmacokinetics
Accumulation ratio (AR) | Day1-15 (MAD)
  Pharmacokinetics
Accumulation ratios for Cmax | Day1-15 (MAD)
  Pharmacokinetics
Accumulation ratios for AUC | Day1-15 (MAD)
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Angela Rowland, Principal Investigator — CMAX Clinical Research Pty Ltd
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: No